CLINICAL TRIAL: NCT00779220
Title: A Randomized, Double-blind, Parallel-group, Study to Evaluate the Efficacy, Safety and PK/PD of Ocrelizumab in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate Therapy
Brief Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics/Pharmacodynamics (PK/PD) of Ocrelizumab in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JA21963
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo; Drug: methotrexate
- 2 (Experimental)
  Interventions: Drug: methotrexate; Drug: ocrelizumabu 50mg
- 3 (Experimental)
  Interventions: Drug: methotrexate; Drug: ocrelizumabu 200mg
- 4: (Experimental)
  Interventions: Drug: methotrexate; Drug: ocrelizumab 500mg

INTERVENTIONS:
Drug: placebo — Intravenous repeating dose
  Arms: 1
Drug: methotrexate — Oral repeating dose
Drug: ocrelizumabu 50mg — Intravenous repeating dose (50mg)
  Arms: 2
Drug: ocrelizumabu 200mg — Intravenous repeating dose (200mg)
  Arms: 3
Drug: ocrelizumab 500mg — Intravenous repeating dose (500mg)
  Arms: 4:

SUMMARY:
This study will evaluate the efficacy, safety and PK/PD of ocrelizumab at each dose in combination with methotrexate（MTX）in patients with active rheumatoid arthritis (RA). The data from this study will also be compared with those from a clinical study of ocrelizumab in patients with active RA that was conducted in the U.S.

DETAILED DESCRIPTION:
This study will evaluate the efficacy, safety and PK/PD of ocrelizumab at each dose in combination with MTX in patients with active RA. The data from this study will also be compared with those from a clinical study of ocrelizumab in patients with active RA that was conducted in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for ≧6 months according to the revised 1987 ACR criteria for the classification of RA.
* Adult patients, ≧20 years of age.
* Receiving methotrexate at a dose of 6 to 8mg/week（oral）for ≧12 weeks, with a stable dose for the last 4 weeks before treatment.
* Positive serum RF.

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA, or Significant systemic involvement secondary to RA (including but not limited to vasculitis, pulmonary fibrosis, or Felty's syndrome).Patients with secondary Sjögren's syndrome or secondary limited cutaneous vasculitis with RA are eligible.
* Functional Class Ⅳ as defined by the ACR Classification of Functional Status in RA.
* History of or current inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease or other overlap syndrome).
* Any surgical procedure (except for minor surgeries requiring local or no anaesthesia and without any complications or sequelae) within 12 weeks prior to or planned within 24 weeks after baseline.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR20 response. | week 24

SECONDARY OUTCOMES:
Percentage of patients with ACR20, 50, and 70 response, and the components of this outcome. | very 4 Weeks, from Week 4 to Week 24
EULAR response rate. | Every 4 Weeks, from Week 4 to Week 24
DAS 28, HAQ-DI score. | Every 4 Weeks, from Week 4 to Week 24
FACIT Fatigue Scale score | Weeks 4,12,and 24
Weeks 4,12,and 24 | Length of study
Incidence of human anti-human(ocrelizumab) antibodies (HAHA) | Length of study
Pharmacokinetics and Pharmacodynamics of ocrelizumab. | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Naritoshi Mochidome, Study Chair — Chugai Pharmaceutical
Locations (7):
- Japan (7):
  - Chugoku region, Chugoku
  - Chubu region, Chūbu
  - Hokkaido Region, Hokkaido
  - Kanto Region, Kanto
  - Kinki Region, Kinki
  - Kyusyu region, Kyusyu
  - Sikoku region, Sikoku

REFERENCES:
- [Derived] Harigai M, Tanaka Y, Maisawa S; JA21963 Study Group. Safety and efficacy of various dosages of ocrelizumab in Japanese patients with rheumatoid arthritis with an inadequate response to methotrexate therapy: a placebo-controlled double-blind parallel-group study. J Rheumatol. 2012 Mar;39(3):486-95. doi: 10.3899/jrheum.110994. Epub 2012 Jan 15. PMID 22247354